CLINICAL TRIAL: NCT02370966
Title: Berry Intake - Effects on Systemic and Oral Inflammation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kristianstad University (Other)
Responsible Party: Principal Investigator, Cecilia Widen, Researcher, Kristianstad University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KristianstadU
Record Dates: First submitted 2015-02-12; First posted 2015-02-25 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Potato starch (Placebo Comparator): Potato powder will be incorporated in the placebo product.
  Interventions: Dietary Supplement: Berry powder
- Berry powder (Active Comparator): Several different berry powders including rose hip, bilberry, blackcurrant, sea buckthorn, and lingonberry will be prepared and studied.
  Interventions: Dietary Supplement: Berry powder

INTERVENTIONS:
Dietary Supplement: Berry powder — Berry and gingivitis trial
  Other Names: Natural berries

SUMMARY:
The purpose of this study is to determine whether intake of berry powder effective in the treatment of systemic and oral inflammation.

DETAILED DESCRIPTION:
Summary About 10-15 % of the adult population in Sweden suffers from periodontitis, which is an inflammatory response to certain oral bacteria. The first stage of periodontitis is termed gingivitis, which is clinically defined by swollen tissue, redness and bleeding in the gingiva. If the inflammatory process could be attenuated, this would greatly reduce the risk of developing periodontitis.

Diet is of importance for the development and prevention of chronic diseases. Berries contain compounds that can act as anti-inflammatory agents and this bioactivity may reduce the risk of disease. A recent meta-analysis of publications in this area revealed a dearth of experimental and clinical data on the impact of berry intake on inflammatory conditions. Studies which detail berry intake/dosage and period of dosage to exert an effect is particularly lacking, in terms of the positive effects of berries on anti-inflammatory conditions. The purpose of this project is to:

* Demonstrate the impact of daily intake of freeze-dried berries on the clinical degree of chronic inflammation by studying changes in the degree of gingivitis.
* To study the presence of pro- and anti-inflammatory markers locally in gingival tissue, saliva and through analysis of serum samples.
* To analyze dose response relationship for different berry powders by investigating clinical and biomedical effect.

Background Many diseases have a significant inflammatory pathogenesis which can be difficult to control. In traditional medicine symptoms and inflammatory processes are treated with pharmaceuticals. Many pharmaceuticals show side-effects that have economic and environmental consequences both for the individual and the environment. It has for centuries been known that plants have anti-inflammatory and healing effects. An early example of how plants came in use for medical treatment is the work of Carl von Linné and his practice as a botanist and physician.

In modern times complimentary alternative medicine has claimed that intake of fruit and berries in different compositions has anti-inflammatory effects. Some of these claims have been difficult to evaluate since studies to highlight anti-inflammatory benefit have often not been well conducted. There is a conspicuous lack of data on clinically effective doses of plant extracts. The Swedish National Food Agency contends that the daily intake of vegetables, fruits and berries should be 500 grams for adults, although few people in Sweden reach these recommendations.

Fruits and berries are not considered pharmaceuticals but are often termed 'nutraceuticals'. Despite a lack of scientific grounds for the medicinal use of fruits and berries, there are today a very large range of health products based on fruits and berries. It is, therefore, of importance to scientifically investigate which fruits and berries that have demonstrable anti-inflammatory effects that is to specifically study biomarkers and clinical conditions with adult individuals. It is also vital to develop a palatable form of administration of the berries that would facilitate regular intake of a naturally based product.

Using biomedicine as a starting point we aim to study anti-inflammatory effects in clinical, randomized, case control, studies. Our primary objective is to treat adult individuals with gingivitis. In general, gingivitis makes up a common chronic condition with adults and it occurs in more than half the population. From a clinical perspective there are well established methods to investigate inflammation in the mouth. The presence of inflammatory biomarkers in the mouth can be conveniently and efficiently measured. Through standard methods for blood sampling one can study the same inflammatory biomarkers and thus analyze which general effects the intake of a test product may have.

Method A daily intake of 500 g is difficult to achieve. Freeze-dried berry powder is a distribution form that would enable regular intake of a naturally based product. We intend to investigate dose-response relationship of different berries, such as bilberries, black currant, lingonberries, rose hip, and sea buckthorn. The selection of berries will be based on accessibility, assumed acceptance and variation of nutrients and commercial conditions. Our earlier studies on bilberries will be used as a reference. All berry powders that will be used in the study will be analyzed for sugar content of micronutrients.

We will analyze clinical effects of the degree of gingivitis and changes of known biomarkers of inflammation in serum, saliva and gingival fluid. We will start with a low dose and double the dose each week. We have made the assumption that the content dry substance in berries is about 10 %, i.e. 50 g freeze-dried berries would correspond to 500 g fresh berries. We will start with 6.25 g berry powder and double the dosage each week until we reach a maximum dosage of 50 g according to the Swedish National Food Agencies recommendations.

The clinical investigations will include a routine dental examination assessing for probing depths at teeth, the extent of gingival bleeding, and presence of plaque accumulation on teeth. Serum, saliva, and gingival fluid samples will be collected to assess for bacteria and cytokine levels. The dental nurse that will conduct the clinical investigation will have no information whether participating individuals have been assigned a berry powder or placebo. Placebo will consist of potato starch. The clinical and biomedical parameters will be studied weekly as seven days is the time required to assure clinical effects and assumed to be sufficient to reach steady-state levels on markers of inflammation. The aim is to identify dose-response relationship and to rank the effects of the different berries.

The examination of biomarkers is based on Luminex Technology. The Luminex system enables analysis of a combination of markers of inflammation in small samples volumes. Our experience from the pilot study has showed that in order to obtain statistical power for VEGF and MIP-1α 16 individuals are required. We plan to include 20 individuals in each series to compensate if some individuals don't complete the study. Inclusion criteria is registration of lingual bleeding on the first and second molar in the lower jaw.

ELIGIBILITY:
Inclusion Criteria:

* minimum of 20 teeth
* bleeding on probing >25 %
* participate in routine dental examinations

Exclusion Criteria:

* on anti-inflammatory medication
* current treatment with antibiotics or intake of antibiotics 3 months before participating in the study
* pregnancy
* smoker
* unwilling to refrain from nutraceuticals during the study period
* unwilling to give detailed information on diet intake during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Changes in the extent of gingivitis, as determined by severity of gingival bleeding, before and after study procedures. | Once a week over five weeks.

SECONDARY OUTCOMES:
Change in levels of vascular endothelial growth factor in serum, saliva and gingival fluid in relation to gingival inflammation, as determined by severity of gingival bleeding, before and after study procedures. | Once a week over five weeks.
Change in levels of vascular endothelial growth factor in serum, saliva and gingival fluid in relation to amount of berry intake before and after study procedures. | Once a week over five weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Rutger Persson, PhD, DDS, Study Director — University of Kristianstad
Locations (1):
- University of Kristianstad, Kristianstad, Skåne County, Sweden